CLINICAL TRIAL: NCT01137331
Title: A Multicenter, Randomised, Double Blind, Placebo-controlled Study of Efficacy, Safety, and Tolerability of Kaprolac® K301 for the Treatment of Seborrhoeic Eczema (SE) of the Scalp
Brief Title: K301 for the Treatment of Seborrhoeic Eczema (SE) of the Scalp
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Moberg Pharma AB (Industry)
Responsible Party: Kjell Rensfeldt MD, Moberg Derma AB
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K301-I
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Last update posted 2010-06-04 (Estimated); Status verified 2010-06

CONDITIONS: Seborrhoeic Eczema of the Scalp
Keywords: seborrhoeic eczema; scalp; dandruff; K301; K40
MeSH Terms: conditions — Dermatitis, Seborrheic; Dandruff

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- K301 (Experimental): K301 applied topically to the affected area of the scalp once daily during the 4 weeks. Treatment is to be applied before bedtime and can be washed out with the patient's normal shampoo in the morning.
  Interventions: Drug: K301
- Placebo (Placebo Comparator): Placebo applied topically to the affected area of the scalp once daily during the 4 weeks. Treatment is to be applied before bedtime and can be washed out with the patient's normal shampoo in the morning.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: K301 — Liquid- applied once daily prior to bed
  Other Names: K40
  Arms: K301
Drug: Placebo — Liquid- applied once daily prior to bed
  Arms: Placebo

SUMMARY:
Seborrhoeic eczema (SE) is a chronic, inflammatory skin disorder confined to areas of the head and trunk where sebaceous glands are most prominent. The severity varies from mild dandruff to exfoliative erythroderma that ranges from mild, patchy scaling to widespread, and thick, adherent crusts. The worldwide prevalence of SE is 3-5%, although dandruff, the mildest form of the disorder affects up to 15-20% of the population.

In this multicentre, randomised, double-blind, placebo-controlled phase III study, adult SE patients are treated once daily for 4 weeks. The population for this study is patients with mild to moderate SE.

The primary endpoint for this study is the efficacy of K301 compared to placebo which was based on the sum score for erythema and desquamation after 4 weeks of daily application. Secondary endpoints are to evaluate safety and tolerability as well as efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (including fertile women)
* 18-70 years of age
* Seborrhoeic eczema of the scalp for at least 2 months
* Presenting erythema and desquamation of mild to moderate intensity
* Signed written informed consent

Exclusion Criteria:

* Seborrhoeic eczema or any other cutaneous disease of the face or scalp requiring a specific topical treatment (corticosteroids, antifungals, selenium sulphide, antibiotics, retinoids, benzoyl peroxide or a-hydroxyacids) during the previous 15 days
* Oral treatment with cyclines, lithium, antifungals or inhaled corticosteroids during the previous month
* Use of systemic corticosteroids and retinoids during the previous 2 months
* Seborrhoeic eczema associated with Parkinson's disease or HIV infection
* Current or any history of ear, nose, and throat carcinoma
* Current or any history of severe concomitant disease according to Investigator's judgement
* Allergy to any of the tested treatment components
* Subject who has been previously enrolled in the phase II study K40-3 investigating Kaprolac® K40

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2008-02; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Erythema and desquamation scores | Week 4
  The sum of erythema and desquamation scores at Week 4

SECONDARY OUTCOMES:
Erythema and desquamation scores | Week 2
  The sum of erythema and desquamation scores at Week 2
Erythema score | Weeks 2 and 4
  Erythema score at Week 2 and 4
Desquamation score | Weeks 2 and 4
  Desquamation score at Week 2 and 4
Investigator's global evaluation | Week 4
  Investigator's global evaluation at Week 4
Patient's global evaluation | Week 4
  Patient's global evaluation at Week 4
Pruritus/burning score | Weeks 2 and 4
  Patient's pruritus/burning score at Week 2 and 4
Dandruff score | Weeks 2 and 4
  Patient's dandruff score at Week 2 and 4
Proportion of responders | Weeks 2 and 4
  Proportion of responders at Week 2 and 4
Adverse events | Weeks 2, 4 and 5
  Adverse events classified by body system and preferred term

CONTACTS AND LOCATIONS:
Overall Officials: Åke Svensson, MD, PhD, Principal Investigator — Hudkliniken UMAS
Locations (19):
- Sweden (19):
  - Läkarhuset Farsta Centrum, Farsta
  - Hedgrindhälsan AB, Gävle
  - Centrumläkarna, Gothenburg
  - Kristinelundskliniken Hudläkarmottagningen, Gothenburg
  - Me3plus clinical trials, Gothenburg
  - Fruängens Läkarhus, Hägersten
  - Hudmottagningen, Helsingborg
  - Familjehälsan, Hofors
  - Din doktor i Stockholm AB, Huddinge
  - Capio Cityklinik, Kristianstad
  - Limhamns Läkargrupp- Tärnan, Limhamn
  - Hudläkarna i Linköping, Linköping
  - Center för Läkemedelsprövningar, Malmo
  - Hudkliniken UMAS, Malmo
  - Möllevångens Husläkargrupp, Malmo
  - Hjortens VC, Trollhättan
  - VC Silentzvägen Praktikertjänst, Uddevalla
  - Hälsojouren, Uppsala
  - Läkarhuset Uppsala, Uppsala